# 18F-AV-1451-A05 SAP Confirmatory Addendum v1.0

An Open Label, Multicenter Study, Evaluating the Safety and Imaging Characteristics of 18F-AV-1451 in Cognitively Healthy Volunteers, Subjects With Mild Cognitive Impairment, and Subjects With Alzheimer's Disease

NCT02016560

Approval date: 05 Jan 2018

# Protocol No. 18F-Flortaucipir-A05

An open label, multicenter study, evaluating the safety and imaging characteristics of flortaucipir in cognitively healthy volunteers, subjects with Mild Cognitive Impairment, and subjects with Alzheimer's Disease

Confirmatory (Second Phase) Addendum to Statistical Analysis Plan

Prepared for: Avid Radiopharmaceuticals, Inc

Final Version 1.0 Date 05Jan2018

Prepared by:

**Chiltern International Inc.** 

## **Revision History**

| Version | Date | Revision Author | Comments |
|---------|-----------|-----------------|----------|
| 1.0 | 05Jan2018 | | |

This document is the confidential information of Avid Radiopharmaceuticals. It may not be disclosed to parties not associated with the clinical investigation or used for any purpose without the prior written consent of Avid Radiopharmaceuticals.

# SIGNATURE PAGE



# **Table of Contents**

| 1 | LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 4 |
|---|---|---|
| 2 | INTRODUCTION | 6 |
| 3 | STUDY OBJECTIVE | 6 |
| 4 | STUDY DESIGN | 6 |
| | 4.1 Blinding | 7 |
| 5 | EFFICACY VARIABLES | |
| | 5.4.1 Quantitative Imaging Assessment of Flortaucipir Scan 5.4.2 Quantitative Imaging Assessment of Florbetapir Scan 5.4.3 Cognitive and Functional Assessments 5.4.4 Volumetric MRI Assessments | 7<br>7 |
| 6 | | |
| | 6.1 GENERAL METHODOLOGY | _ |
| 7 | STATISTICAL ANALYSIS | 8 |
| | 7.1 DISPOSITION OF SUBJECTS | 8<br>8 |
| | Measurement | 9 |
| | 7.3.3 Relationship between Quantitative Tau Load and Other Biomarkers | 9 |
| 8 | COMPUTER SOFTWARE | 9 |
| 9 | REFERENCES | 9 |

# 1 LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

**Table 1: Abbreviations and Definitions of Terms** 

| 1.0 | 1:10 |
|----------------|------------------------------------------------|
| Αβ | amyloid-β |
| AD | Alzheimer's disease |
| ADAS-Cog | Alzheimer's Disease Assessment Scale-Cognitive |
| AE | adverse event |
| ANART | American National Adult Reading Test |
| ATC | Anatomical Therapeutic Chemical |
| BMI | body mass index |
| BNT | Boston Naming Test |
| C | Celsius |
| cm | centimeters |
| CNS | central nervous system |
| CRF | case report form |
| CRO | contract research organization |
| CSF | cerebrospinal fluid |
| DBP | diastolic blood pressure |
| DSST | digit symbol substitution test |
| ECG | electrocardiogram |
| EDTA | ethylenediaminetetraacetic acid |
| eCRF | electronic case report form |
| FAQ | Pfeffer Functional Activities Questionnaire |
| FDG | <sup>18</sup> F- flurodeoxyglucose |
| Н | high |
| hCG | human chorionic gonadotropin |
| IND | investigational new drug |
| IV | intravenous |
| JOLO | Benton Judgment of Line Orientation Test |
| K <sub>d</sub> | dissociation constant |
| kg | kilograms |
| L | low |
| LOC | loss of consciousness |
| LS | least squares |
| max | maximum |
| MBq | megabecquerel |
| mCi | millicuries |
| MCI | mild cognitive impairment |
| MedDRA | Medical Dictionary for Regulatory Activities |
| min | minimum |
| l . | l |

| ) (I) (I)) ( | |
|---|---|
| MMRM | mixed model repeated measures |
| MMSE | Mini-Mental State Examination |
| MRI | magnetic resonance imaging |
| mSv | millisievert |
| n | number of subjects |
| N | normal |
| nM | nanomolar |
| OSU TBI-ID | Ohio State University Traumatic Brain Injury Identification Method |
| PET | positron emission tomography |
| ROI | region of interest |
| RR | respiration rate |
| SAP | statistical analysis plan |
| SBP | systolic blood pressure |
| SD | standard deviation |
| SOC | system organ class |
| SOP | standard operating procedure |
| SUVr | standardized uptake value ratio |
| TBI | Traumatic Brain Injury |
| TEAE | treatment-emergent adverse event |
| TEMP | temperature |
| WHO | World Health Organization |

#### 2 INTRODUCTION

The quantitative assessment of Flortaucipir scan (standard uptake value ratio, SUVr) is important in helping to better understanding how brain tau load (as measured by flortaucipir scans) correlates with cognitive function progress. However quantitative analysis of tau PET imaging is a rapidly evolving field and not yet routine in Core laboratories. Therefore, Avid's imaging science team will assume the role for this part of imaging analysis, and the results (SUVr values) will be used in exploratory analyses in this study, and will be reported in CSR with other analysis results. To keep Avid staff blinded to the key information, the quantitative scan analysis process will be happening post main study database lock, which including the lock of both clinical and tau/amyloid imaging scan qualitative assessments (visual reads) results. Therefore this addendum SAP is created to describe the relative steps, and the planned analyses that will include imaging quantitative assessments.

#### 3 STUDY OBJECTIVE

This SAP will detail the exploratory analyses that involve flortaucipir and florbetapir quantitative assessments. All the analyses included here are for exploratory purpose.

#### 4 STUDY DESIGN

The process of imaging quantitative analysis (including both flortaucipir and florbetapir imaging) will be following the steps as below:

Database lock at TPO as scheduled, inlcuding imaging visual reads for both flortaucipir and florbetapir (which will all happen with the independent imaging core lab), and clinical data collection/cleaining Once DBL is completed, the imaging TPO will start to transfer flortaucipir and florbetapir scans to Avid. The Avid imaging science team will start to analyze scans quantitatively once the scans are in place. During this analysis process, Avid imaging science team will remain blinded to clinical and visual read data

Once the Avid imaging team finished the quantitative analysis, quantitative assessment data (SUVr values) will be transferred to TPO for addendum TLF production, following the analyses as detailed in this addendum

The details of this process is documented in A05 study blinding document.

# 4.1 Blinding

Avid imaging science team will assume the role of quantitative imaging analyses, including both flortaucipir scans, and florbetapir scans. Therefore the team will be blinded to any other study data, including both clinical and imaging qualitative assessments until the analyses results are sent to TPO for addendum TFL production, and addendum lock memo signed.

#### 5 EFFICACY VARIABLES

#### 5.1.1 Quantitative Imaging Assessment of Flortaucipir Scan

For the flortaucipir image, standardized uptake value ratios (SUVr) will be calculated using a subject specific white matter based parametrically derived reference region (parametric estimate of reference signal intensity, PERSI¹). The global cortical target ROI will consist of a weighted average of voxels found, through multi-block barycentric discriminant analysis (MUBADA) to best sepaparate the amyloid positive AD/MCI and amyloid negative CN subjects, from the A05 exploratory cohort. In addition, cortical region ROI SUVr based on modified AAL regions will also be calculated. The details are documented in imaging analysis plan.

## 5.1.2 Quantitative Imaging Assessment of Florbetapir Scan

For the Florebetapir 18 F image, standardized uptake values (SUV) for target areas such as the frontal cortex, temporal cortex, parietal cortex, posterior cingulate cortex, anterior cingulate cortex and the precuneus will be calculated from each image. Standardized uptake value ratios (SUVr) will be calculated for target areas by calculating the ratio of the specific SUV to the entire cerebellum SUV. The global cortical average SUVr will be calculated as the average across these six target brain regions.

#### 5.1.3 Cognitive and Functional Assessments

Cognitive and functional assessments as detailed in section 6.4.2.2 of A05 confirmatory SAP, include MMSE, ADAS, FAQ, and CDR.

# 5.1.4 Volumetric MRI Assessments

Volumetric MRI assessments are detailed in section 6.4.2.6 of A05 confirmatory SAP.

#### 6 STATISTICAL METHODS

# 6.1 General Methodology

Frequency distributions including counts and percentages will be included for all categorical outcomes. Summary statistics including mean, standard deviation, median, minimum and maximum values will be presented for all continuous outcomes. Unless otherwise specified, hypothesis testing will be two-sided with type I error rate of 0.05.

All statistical analyses will be performed using SAS® version 9.3 or higher.

# 6.2 Adjustments for Covariates

None.

#### 7 STATISTICAL ANALYSIS

# 7.1 Disposition of Subjects

Flortaucipir and florbetapir images that are not quantifiable due to reasons such as technical issues and etc. will be documented in details in a note to file (NTF). The number of subjects with imaging received by Avid imaging science team, number of subjects with imaging quantitative analysis completed, and number of subjects with imaging scans fail to complete quantitation will be presented in a table, along with reasons of why quantitation failed. A listing will also be provided.

# 7.2 Analysis Populations

## 7.2.5 Efficacy Population

The efficacy population for the analyses covered in this addendum SAP will include all subjects with a valid flortaucipir quantitative scan analysis result (SUVr value).

## 7.3 Analysis of Efficacy Parameters

# 7.3.1 Relationship between Quantitative Tau Load and Baseline Cognitive/Functional Measurement

To evaluate the relationships between brain tau load as measured by flortaucipir SUVr value and the cognitive and functional assessments, scatter plots between MUBADA SUVr and each of the baseline cognitive and functional assessments as detailed in section 5.1.3 will be generated. Pearson correlation analyses will be conducted for each of these pairs, and the correlation coefficient will be provided along with the 95% confidence intervals (CI), and the associated p-values.

# 7.3.2 Relationship between Quantitative Tau Load and Cognitive/Functional Change at 18 Months Visit

Similar analyses will be conducted as detailed in section 7.3.1, by changing baseline cognitive/function measurements to cognitive/functional measurements change from baseline at 18 months.

# 7.3.3 Relationship between Quantitative Tau Load and Other Biomarkers

Similar analyses will be conducted as detailed in section 7.3.1, by changing baseline cognitive/function measurements to the biomarkers such as below:

- 1. Amyloid level as assessed by florbetapir SUVr;
- 2. MRI volumetric assessments as detailed in A05 confirmatory SAP section 6.4.2.6.

#### 8 COMPUTER SOFTWARE

All analyses will be performed by Chiltern International Inc. using Version 9.3 or later of SAS® software. All summary tables and data listings will be prepared utilizing SAS® software.

For continuous variables, descriptive statistics (number of subjects [n], mean, standard deviation [SD], median, minimum, maximum, 25<sup>th</sup> pct, and 75<sup>th</sup> pct) will be generated. The standard operating procedures (SOPs) of Chiltern International Inc. will be followed in the creation and quality control of all data displays and analyses.

#### 9 REFERENCES

 Southekal S, Devous MD, Kennedy I, Navitsky M, Lu M, Joshi AD, Pontecorvo MJ, Mintun MA. Flortaucipir F 18 Quantitation using a Parametric Estimate of Reference Signal Intensity (PERSI). Journal of Nuclear Medicine (submitted).